CLINICAL TRIAL: NCT07048860
Title: A ICOPE Intense Program Combined With Ketone Ester Pilot Study
Brief Title: ICOPE INTENSE-K Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/24/0519; 2025-A00891-48 (Other: ANSM)
Record Dates: First submitted 2024-12-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ageing
Keywords: cognition; morbility; intrinsic capacity; biomarker of aging
MeSH Terms: interventions — Dietary Supplements; Cholecalciferol; Docosahexaenoic Acids; Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICOPE-intense group (Experimental): ICOPE intense intervention + placebo
  Interventions: Other: ICOPE intense intervention; Dietary Supplement: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: OMega 3; Dietary Supplement: vitamin B9; Dietary Supplement: Vitamin B12; Dietary Supplement: Leucin-rich whey
- The ICOPE-intense + Ketone Ester (KE) group (Experimental): ICOPE intense intervention + nutritional ketone esther suplementation
  Interventions: Other: ICOPE intense intervention; Dietary Supplement: Ketone Ester (KE) supplementation; Dietary Supplement: Vitamin D3; Dietary Supplement: OMega 3; Dietary Supplement: vitamin B9; Dietary Supplement: Vitamin B12; Dietary Supplement: Leucin-rich whey
- The Ketone group (Experimental): Usual ICOPE step 1 + ketone esther supplementation
  Interventions: Dietary Supplement: Ketone Ester (KE) supplementation; Other: ICOPE Step 1
- Control group (Placebo Comparator): Usual ICOPE step 1 + placebo
  Interventions: Dietary Supplement: Placebo; Other: ICOPE Step 1

INTERVENTIONS:
Other: ICOPE intense intervention — The ICOPE-intense intervention (45 hours centre-based (in-group and in-person) multidomain intervention, everyday home-based lifestyle improvement, and weekly individual phone/video call for support)
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Dietary Supplement: Ketone Ester (KE) supplementation — 12.5g once a day of KE for week 1, and 25g once a day of KE supplementation week 2 to week 8.
  Arms: The ICOPE-intense + Ketone Ester (KE) group; The Ketone group
Dietary Supplement: Placebo — 2.5 g of nonketogenic canola oil
  Arms: Control group; ICOPE-intense group
Dietary Supplement: Vitamin D3 — 2 sprays (i.e. 2000 iu) per day in the morning for 60 days
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Dietary Supplement: OMega 3 — 1000 mg: 1 table per day in the morning during 60 days
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Dietary Supplement: vitamin B9 — 5 mg cp: 1 tablet morning and 1 tablet evening for 60 days
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Dietary Supplement: Vitamin B12 — 250 microgram: 1 tablet per day in the morning for 30 days, then 1 tablet every 10 days for 30 days
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Dietary Supplement: Leucin-rich whey — In case of Sarcopenia or low protein intake (<1.2 g/kg/day), Oral Nutritional Supplementation enriched in essential amino acid (leucin)
  Arms: ICOPE-intense group; The ICOPE-intense + Ketone Ester (KE) group
Other: ICOPE Step 1 — usual ICOPE Step 1
  Arms: Control group; The Ketone group

SUMMARY:
ICOPE could constitute the reference model of care for healthy aging. More specifically, our hypothesis is that the intervention implemented in ICOPE may directly or indirectly prevent immuno-senescence, the loss of mobility and the cognitive decline. In future Geroscience clinical trials, ICOPE-Intense could become a benchmark to reduce the rate of aging with a strong non-pharmacological intervention and state a reference intervention to compare with new gerotherapeutic drugs.

DETAILED DESCRIPTION:
In this pilot study, the concept of prevention proposed by the WHO, for everyday life is taken to the extreme to be able to judge what is the maximum effect size on key functions of aging (mobility, cognition, immunity) that can be expected and achieved by a nonpharmacological intervention. The results obtained will constitute reference data for the future, during the investigation on new gerotherapeutic drugs or other nonpharmacological interventions. Taking into account the hypothesis of a synergistic effect between Ketones and non-pharmacological intervention, the intense ICOPE program makes it possible to study the effect size of Ketones under optimal experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Independent-living (ADL ≥5/6)
* Men and women
* Mobility impairment (5 Chair-rise test >12 seconds)
* Sedentarism (spend six or more hours per day sitting or lying down)
* Positive screening for cognitive impairment according to the ICOPE screening tool with MMSE [25-28]
* BMI ≥25 kg/m2

Exclusion Criteria:

* Unintentional weight loss (≥10%) in past 6 months
* Dementia
* Life-threatening illnesses, with a life expectancy (judged by the investigating doctor) of less than 1 year
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina or any other contraindication to physical activity (as determined by a physician) or comorbid disease that would impair ability to participate in the ICOPE intense intervention such as renal failure on hemodialysis, severe psychiatric disorder (depressive participant will not be excluded)
* Organizational inability (three-time per week during the 60 days)
* Living in a Nursing-Home
* Under legal protection measure (guardianship, curatorship, safeguard of justice

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of the effect size of the intervention on the cognitive function | 60 days
  The cognitive function will be assessed using the Cambridge Neuropsychological Test Automated Battery (CANTAB), a computerized neuropsychological test with a game-like and non-verbal environment that assesses the different cognitive domains, at baseline and day 60.
Estimation of the effect size of the intervention on the muscle function | 60 days
  The muscle function will be assessed using 3 validated clinical approaches that investigate muscle endurance, muscle strength/power and muscle mass at baseline and day 60:
  * Muscle endurance will be tested using the 6-min walk test
  * Lower body power assessed with the 5-time chair rise test
  * Muscle mass will be assessed using the Deuterated-Creatine Dilution approach
Estimation of the effect size of the intervention on the immune function | 60 days
  The analysis of immune function will be determined by the analysis of PBMC collected and bio banked at baseline and at 60 days. Specific assay decisions will be determined and fixed in 2026 by the scientific adversary board of the financer application.

CONTACTS AND LOCATIONS:
Locations (1):
- Cité de la santé - Hopital La Grave, Toulouse, France